CLINICAL TRIAL: NCT03349372
Title: Impact of Systematic Pulmonary Follow-up After Hematopoietic Stem Cell Transplantation
Brief Title: Impact of Pulmonary Follow-up After Stem Cell Graft
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_007
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — Hematopoietic stem cell transplantation

SUMMARY:
Allogeneic hematopoietic stem cell transplantation is the only possible treatment for many malignant and non-malignant hemopathies. The graft-versus-host immunological reaction (GvH) is a frequent and sometimes serious complication. The objective is to study whether a systematic and early follow-up by a lung specialist of allografted patients would allow an earlier diagnosis of GvH with pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* patients with a hematopoietic stem cell transplantation

Exclusion Criteria:

* Death within 100 days post-surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients from Hospices Civils de Lyon, Lyon, France with blood cancer undergoing a hematopoietic stem cell transplantation between January 2013 and July 2016
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Medical complications | Medical complications, especially Graft-versus-Host reaction with pulmonary complications occurring within 100 days post-surgery are studied
  100 days after allograft

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No